CLINICAL TRIAL: NCT06686550
Title: The Impact of Preoperative Sleep Disorders on the Incidence of Postoperative Delirium in Children Undergoing Congenital Heart Surgery: A Prospective, Observational, Cohort Study
Brief Title: Preoperative Sleep Disorders and Postoperative Delirium in Children Undergoing Congenital Heart Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Yan Fuxia (Other)
Responsible Party: Sponsor-Investigator, Yan Fuxia, Chinese Academy of Medical Sciences, Fuwai Hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Other Study IDs: 2024-2414
Record Dates: First submitted 2024-10-31; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Delirium - Postoperative; Sleep Problems; Congenital Heart Disease (CHD)
MeSH Terms: conditions — Emergence Delirium; Parasomnias; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children scheduled to undergo elective congenital heart disease repair surgery with CPB
  Interventions: Other: This is a observational study and there is no intervention.

INTERVENTIONS:
Other: This is a observational study and there is no intervention. — This is a observational study and there is no intervention.

SUMMARY:
The investigators are going to conduct a prospective observational cohort study in pediatric patients aged 28 days to 14 years old scheduled for elective cardiac surgery with cardiopulmonary bypass. The primary purpose of this study is to explore the effect of preoperative sleep disturbance on the incidence of postoperative delirium. Sleep status will be assessed using the Brief Infant Sleep Questionnaire(BISQ) and Children's Sleep Habits Questionnaire (CSHQ), and postoperative delirium status will be evaluated by Cornell assessment of pediatric delirium(CAPD). During the peri-operative period, children will wear actigraphs to record their sleep parameters.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 28 days and less than 14 years old；
* Scheduled to undergo elective corrective surgery for congenital heart disease under cardiopulmonary bypass.

Exclusion Criteria:

* Emergency surgery;
* Combined with severe hepatic and renal dysfunction (with a diagnosis of acute or chronic renal insufficiency or requiring renal replacement therapy; with a diagnosis of acute or chronic hepatic insufficiency or requiring artificial liver treatment);
* Combined with non-cardiac malformations (adenoidal hypertrophy, tracheobronchial stenosis and ocular disorders);
* History of preoperative cerebral ischemia or haemorrhage;
* Refuse to sign the informed consent form or the child has poor compliance.

Ages: 28 Days to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged more than 28 days and less than 14 years old who are scheduled to undergo elective corrective surgery for congenital heart disease under cardiopulmonary bypass.
Sampling Method: Probability Sample
Enrollment: 435 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium | Postoperative 7 days

SECONDARY OUTCOMES:
The proportions of subtypes of postoperative delirium( hypoactive, hyperactive, and mixed). | Postoperative 7 days
Pain defined by the Face, Legs, Activity, Cry, and Consolability scale | Postoperative 7 days
  The FLACC scale is a simple and effective tool used to assess pain in infants and non-verbal patients. It stands for Face, Legs, Activity, Cry, and Consolability. Each of these five items is scored on a scale of 0 to 2, with a higher score indicating a greater degree of pain. The total FLACC score, ranging from 0 to 10, provides a quick and reliable assessment of the patient's pain level.
The incidence of postoperative Acute kidney injury | Within postoperative 7 days.
Pulmonary complication | Postoperative 7 days
The incidence of postoperative Liver dysfunction | Postoperative 7 days
The duration of postoperative mechanical ventilation | From the end of the surgery to discharge from the hospital，up to 30 days.
  The total hours needing mechanical ventilation support
The length of intensive care unit stay | From the end of the surgery to discharge from the hospital, up to 30 days.
  The time spent in the intensive care unit.
The length of postoperative hospital stay | From the end of the surgery to the day of discharge from the hospital, up to 30 days..

OTHER OUTCOMES:
Concentration of plasma intestinal injury markers | Before surgery and 24 hours after surgery
  Intestinal fatty acid binding protein, Zonulin, Lipopolysaccharide and so on.
Concentration of plasma blood-brain barrier injury markers | Before surgery and 24 hours after surgery
Concentration of plasma inflammatory factors. | Before surgery and 24 hours after surgery
  The inflammatory cytokines include IL-6，TNF-α，IL-1β，IFN-γ，IL-17, C-reactive protein.
Types and total dosages of sedative and analgesic medications | From the start of the surgery to discharge from the hospital, up to 30 days.